CLINICAL TRIAL: NCT03576235
Title: Safety and Efficacy of PG102P for the coNtrol of prUritus in Patients underGoing Hemodialysis (SNUG Trial): Study Protocol for a Randomized Control Trial
Brief Title: Safety and Efficacy of PG102P for Uremic Pruritus in HD Patients
Acronym: SNUG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Boramae Hospital (Other)
Collaborators: Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); Ewha Womans University Mokdong Hospital (Other); Severance Hospital (Other); Chungnam National University Hospital (Other); Gachon University Gil Medical Center (Other); Kyungpook National University Hospital (Other); DongGuk University (Other)
Responsible Party: Principal Investigator, Chun Soo Lim, Professor, Seoul National University Boramae Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VM_PG102P
Record Dates: First submitted 2018-06-21; First posted 2018-07-03 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Uremic Pruritus
Keywords: Uremic pruritus; Hemodialysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- a treatment group (Experimental): PG102P 1.5 g/day
  Interventions: Drug: PG102P
- a control group (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PG102P — Daily dose of 1.5g
  Arms: a treatment group
Drug: Placebo — Daily dose of placebo
  Arms: a control group

SUMMARY:
In this study (SNUG trial), the investigators aim to investigate the anti-pruritic effect of PG102P in comparison with placebo in 80 patients undergoing HD.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled trial in which one group will be treated with PG102P (1.5 g/day) and the other with a placebo. It is an investigator-initiated clinical trial. A superiority trial is planned to test the hypothesis that PG102P is effective in relieving pruritus for patients with ESRD undergoing HD.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 19 years
2. Patients with adequate HD (Kt/V > 1.2)
3. Maintenance patients undergoing HD with chronic pruritus
4. Mean visual analog scale (VAS) over 4 of the last 5 days in the 14-day pre-observation period
5. Participants who allowed to continue the anti-pruritic drug treatment at the same dosage and administration schedule as used at baseline throughout the study period
6. Patients who agreed to participate in this trial and had written an informed consent

Exclusion Criteria:

1. Intact parathyroid hormone (iPTH) > 1000 pg/mL within 1 month
2. Serum potassium > 7.0 mg/dL
3. HIV Ab (+)
4. Aspartate transaminase (AST) (glutamic oxaloacetic transaminase) or alanine transaminase (ALT) (glutamic pyruvic transaminase) > 3 times the upper limit of normal
5. Scheduled to have kidney transplantation within 3 months
6. Cancer history with current treatment
7. Active infection with current treatment
8. Current itching with dermatologic diseases other than uremic pruritus
9. Pregnancy, childbearing potential during the study period, or breastfeeding
10. Allergy or hypersensitivity reaction to PG102P
11. History of participating another clinical trial within 2 months or planning to participate another clinical trial
12. Not eligible to participate this trial as researchers' decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
VAS change from baseline | the change in VAS between visit 2 (week 0) and visits 3, 4, 5, and 6 (weeks 2, 4, 8, 10)
  The primary endpoint is the change in VAS

SECONDARY OUTCOMES:
serum total IgE | week 0, week 8
  immunoglobulin E
blood Eosinophil count | week 0, week 8
  Eosinophil count
serum ECP | week 0, week 8
  Eosinophil Cationic Protein
serum Ca | week 0, week 8
  serum Calcium
serum P | week 0, week 8
  serum Phosphorus,
serum K | week 0, week 8
  serum Potassium
serum iPTH | week 0, week 8
  intact parathyroid hormone
Questionnaire #1 (KDQOL, Kidney Disease and Quality of Life) | week 0, week 8
  The KDQOL-SF 1.3 includes 43 kidney disease targeted items as well as 36 items that provide a generic core and a overall health rating items (SF-36). The lowest and highest scores of each items are set at 0 to 100, with higher scores reflecting better quality of life.
  1. Kidney disease targeted (number of items)
     Symptoms/Problems (12), Effects of kidney disease (8), Burden of kidney disease (4), Work status (2), Cognitive function (3), Quality of social interaction (3), Sexual function (2), Sleep (4), Social support (2), Dialysis staff encouragement (2), Patient satisfaction rating (1), Overall heath rating (1)
  2. SF-36 (number of items)
  Physical functioning (10), Role-physical (4), Bodily pain (2), General health (5), Mental health (5), Role-emotional (3), Social functioning (2), Vitality (4)
Questionnaire #2 (BDI, Beck's Depression Inventory) | week 0, week 8
  The Beck Depression Inventory (BDI-II) is a 21-question multiple-choice self-report inventory, one of the most widely used psychometric tests for measuring the severity of depression. Each answer is scored 0-3 with a maximum score of 63 points, and higher total scores indicate more severe depressive symptoms.
  0-13: minimal depression, 14-19: mild depression, 20-28: moderate depression, 29-63: severe depression.
serum IL-31 | week 0, week 8
  inflammatory cytokine

CONTACTS AND LOCATIONS:
Overall Officials: Chun Soo Lim, MD, PhD, Principal Investigator — Seoul National University Boramae Medical Center, Seoul, Republic of Korea.
Locations (1):
- Seoul National University Boramae Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Hercz D, Jiang SH, Webster AC. Interventions for itch in people with advanced chronic kidney disease. Cochrane Database Syst Rev. 2020 Dec 7;12(12):CD011393. doi: 10.1002/14651858.CD011393.pub2. PMID 33283264
- [Derived] Kim YC, Park JY, Oh S, Cho JH, Chang JH, Choi DE, Park JT, Lee JP, Kim S, Kim DK, Ryu DR, Lim CS. Safety and efficacy of PG102P for the control of pruritus in patients undergoing hemodialysis (SNUG trial): study protocol for a randomized controlled trial. Trials. 2019 Nov 28;20(1):651. doi: 10.1186/s13063-019-3753-1. PMID 31779697